CLINICAL TRIAL: NCT04214496
Title: Electroencephalographic Biomarker to Predict the Development of Acute Post-operatory Cognitive Dysfunction States: a Protocol of an Observational Study in a Cohort of Patients From Two Centers
Brief Title: Electroencephalographic Biomarker to Predict Acute Post-operatory Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, José Ignacio Egaña Tomic, Director, University of Chile
Other Study IDs: ID19I10345
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Dysfunction; Postoperative Delirium
Keywords: Delirium; Postoperative Delirium; Postoperative Subsyndromal Delirium; Biomarker
MeSH Terms: conditions — Cognitive Dysfunction; Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Postoperative Delirium Risk Patients: Preoperative cognitive function testing- EEG monitorization during surgery - Postoperative function testing
  Interventions: Device: Sedline

INTERVENTIONS:
Device: Sedline — Intraoperative EEG monitorization

SUMMARY:
Acute post-operatory cognitive dysfunction states are one of the most important complications in older patients after surgery. Two acute cognitive dysfunctions have been described: postoperative delirium (PD) and postoperative subsyndromal delirium (PSSD). Patients who develop delirium, both as a complete or incomplete syndrome, have poor long-term outcomes, such as longer length of hospital stay, institutionalization at discharge, and even higher mortality, and consequently, the human and economic costs significantly increase for the health system. Here the research team will use an observational cohort, investigator blinded in two-center with a primary endpoint to validate the relative alpha power ratio as a predictive biomarker of postoperative cognitive dysfunctions.

DETAILED DESCRIPTION:
Acute post-operatory cognitive dysfunction states are one of the most important complications in older patients after surgery. Two acute cognitive dysfunctions have been described: postoperative delirium (PD) and postoperative subsyndromal delirium (PSSD). In previous reports, the incidence of PD in older patients is between 10% to 30%, while PSSD is more frequent 30% to 50%. Patients who develop delirium, both as a complete or incomplete syndrome, have poorer long-term outcomes, such as longer length of hospital stay, institutionalization at discharge, and even higher mortality, and consequently, the human and economic costs significantly increase for the health system.

An early diagnostic and prevention of delirium are the key points to decrease the poor long-term outcomes and health costs. The diagnosis requires cognitive testing to elucidate functional patients' status before and after surgery. The need for a biomarker that may predict the occurrence of PD and PSSD and allow the selection of patients who need prevention strategies is a primary research field.

Here the research team will use an observational cohort, investigator blinded in two-center with a primary endpoint to validate the relative alpha power ratio as a predictive biomarker of postoperative cognitive dysfunctions.

To calculate the sample size, the investigators used values obtained from a previous work in a cohort of 30 patients and decided to compare the prediction ability of MoCA and alpha power ratio. ROC curves and their AUC were used to calculate the prediction ability of MoCA and alpha power ratio. Thus, a sample size of 425 patients was calculated considering an AUC of MoCA = 0.786 and AUC of alpha power = 0.895, a two-tailed test, an alpha error of 0.05 and a power of 0.8 and considering a 25% loss. Investigators consider this study as a pilot validation trial to establish the utility and the capacity of the EEG biomarker for predicting PD and PSSD, the research team aims to include the 25% of the total sample. This yields the need for 106 patients for this preliminary trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Scheduled for high-risk elective surgery
* Need for at least 3 days of hospital stay
* Surgery performed under general anesthesia
* Written informed consent for participation in the trial

Exclusion Criteria:

* Patients with preoperative delirium or dementia
* Patients using neuroleptics drug during the past 6 months
* Patients with a history of encephalopathy, psychosis, stroke or brain trauma with neurologic sequels
* The use of ketamine or dexmedetomidine during surgery
* Emergency surgery
* Mechanical ventilation during the 72 after surgery
* Analphabetism
* Patients who do not talk Spanish
* Patients included in another clinical trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at risk of delirium or subsyndromal delirium after High-risk Surgery will be evaluated in the pre and postoperative period for cognitive dysfunction and the appearance of delirium syndromes. In the intraoperative period, an EEG-based monitorization will be performed using a SedLine (Masimo, CA) Monitor.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Delirium and Subsyndromal Delirium | 5 Postoperative days
  Incidence of Delirium and Subsyndromal Delirium in the cohort

SECONDARY OUTCOMES:
Death | Perioperative period
  Number of deceased patients
Delirium Severity | 5 Postoperative days
  Delirium severity assessed by Cognitive Assessment Method - Severity
Delirium Duration | Perioperative period
  Duration of delirium during the perioperative period
Need for Mechanical Ventilation assistance | Perioperative period
  Number of patients that needed mechanical ventilation
Reintervention | Perioperative period
  Number of patients that needed another surgery after primary intervention
Unanticipated ICU hospitalization | Perioperative period
  Number of patients that needed unanticipated intensive care unit (ICU) care

CONTACTS AND LOCATIONS:
Overall Officials: José I. Egaña, M.D./Ph.D., Study Chair — University of Chile
Locations (2):
- Chile (2):
  - Hospital Clinico Universidad de Chile, Santiago
  - Instituto Nacional del Cancer, Santiago

IPD SHARING:
Plan to Share IPD: Undecided